## Study protocol

Title: From short-term surgical missions towards sustainable partnerships

A survey among members of foreign teams and local doctors

involved in surgical missions.

Study Protocol number: 2019-05

Date of protocol approval: May 15<sup>th</sup> 2019, by the board of Global Surgery Amsterdam

Study type: Survey

The content of the survey is provided below in this study protocol

Initiating organization: Global Surgery Amsterdam (GSA)

www.globalsurgeryamsterdam.com

Collaborating organization: ICOPLAST

www.icoplast.org

General information: Particularly in low- and middle-income countries (LMICs), surgical

missions are conducted on a large scale to provide surgical care. Annually, an estimated 313 million US dollars is spent on surgical missions. Typical missions are short-term, lasting up to several weeks. However, currently we know very little about the actual impact of these missions, including patient outcomes and strategies to make

missions more sustainable.

Therefore we developed an online survey. It is a first step in identifying what is currently being done and what should be done according to the respondent's experiences. The answers are used to provide more clarity on today's practices of short-term missions and

to provide recommendations for the future.

The survey consists of 21 questions. Outcomes will be anonymized.

Participants: Members of foreign teams and local doctors involved in surgical

missions.

Start of distribution: June 2019, by email within the network of GSA and ICOPLAST

End of enrollment: October 2019

Ethical clearance: Not required for this study type



A survey for international and local team members involved in surgical missions in LMICs. Developed by ICOPLAST and Global Surgery Amsterdam

<u>www.icoplast.org</u> www.globalsurgeryamsterdam.com

## Background:

We all aim for improving outcomes of our patients all around the globe. Many of our patients suffer from conditions that can be treated with (reconstructive) surgery. Particularly in low- and middle-income countries, surgical missions are conducted on a large scale to provide this type of care. Annually, an estimated 313 million US dollars is spent on surgical missions. Typical missions are short-term, lasting up to several weeks.

However, currently we know very little about the actual impact of these missions, including patient outcomes and future strategies (Hendriks et al., 2019).

Therefore we developed this questionnaire. It is a first step in identifying what is currently being done and what should be done, according to your valuable experiences in the field. Your data is used to provide more clarity on today's practices of short-term missions.

The questionnaire consists of 21 questions. Please select one answer, and further clarify in the comment box if applicable.

Note: we may ask additional questions in the future if you approve us to contact you. Outcomes will be anonymized.

| Your function * |
|----------------------------------------------------|
| Nurse / physician assistant (Please specify below) |
| Plastic surgeon |
| Orthopedic surgeon |
| General surgeon |
| Other surgeon (Please specify below) |
| Policy officer NGO (Please specify below) |
| Board member NGO |
| Other |
| Q1. Name * Short answer text |
| Q2. Age: * Short answer text |
| Q3. Sex: * Short answer text |
| Q4. Email address: * Short answer text |
| Q5. Nationality: * |
| Short answer text |

| Q6. How many missions did you perform in your life? * |
|---------------------------------------------------------------|
| Short answer text |
| Q7. Country where you performed your last surgical mission: * |
| Short answer text |
| Q8. Name of the hospital and town: * |
| Short answer text |
| Q9. Name of the NGO that supported this mission: * |
| Short answer text |
| Q10. Country where this NGO is based: * |
| Short answer text |

Q11. Please give points over the following potential activities of a visiting team (more points means a more important activity) \*

| | 1 point | 2 points | 3 points | 4 points |
|---|---|---|---|---|
| Provide surgical equipment and consumables for the local team, also for use after the mission left | 0 | 0 | 0 | 0 |
| Provide free treatments | 0 | 0 | 0 | 0 |
| Treat patients yourself | 0 | 0 | 0 | 0 |
| Facilitate<br>teaching of local<br>staff (doctors<br>and/or nurses) | 0 | 0 | 0 | 0 |
| Q12. Is there, in your opinion, an activity missing in question 11? (please explain what activity is important and why) Long answer text | | | | |
| Q13. Should medical registration in the host country be required for specialists performing short-term surgical missions? | | | | |
| Strongly agree | | | | |
| Agree | | | | |
| Neither agree or di | sagree | | | |
| Disagree | | | | |
| Strongly disagree | | | | |

| Comments: |
|---|
| Long answer text |
| Q14. When medical registration was required for your last mission, the process to obtain the documents was straightforward. |
| Strongly agree |
| ○ Agree |
| Neither agree or disagree |
| O Disagree |
| Strongly disagree |
| Comments: |
| Long answer text |
| Q15. What can you say about the collaboration between authorities in LMICs (like the Ministry of * Health, the district health management or the national surgical society) and visiting surgical teams? |
| There is no collaboration and it should be developed as a priority |
| Collaboration is present but improvement is needed |
| Collaboration has no benefits nor disadvantages |
| Collaboration will likely be more harmful than beneficial for the mission |
| Comments: |
| Long answer text |

| Q16. What should have a higher priority in the hospital of your last mission? Teaching in anesthesia care or teaching in surgical care? |
|---|
| Anesthesia care |
| Reconstructive care |
| General surgical care |
| Other surgical care (please specifiy in comments) |
| Comments: |
| Long answer text |
| Q17. A structured follow-up strategy (>6 months) of patients is required for short-term surgical missions. |
| missions. |
| missions. Strongly agree |
| missions. Strongly agree Agree |
| missions. Strongly agree Agree Neither agree nor disagree |
| missions. Strongly agree Agree Neither agree nor disagree Disagree |

| Q18. One month after the mission, an official report on the outcome including all complications *encountered is recommended for all surgical missions. |
|---|
| O Strongly agree |
| ○ Agree |
| Neither agree nor disagree |
| O Disagree |
| Strongly disagree |
| Comments: |
| Long answer text |
| Q19. A written long-term strategy (>5 years) with clear goals, developed by the visiting team and * the local actors together, is recommended at the start of a new project. |
| Strongly agree |
| ○ Agree |
| Neither agree nor disagree |
| O Disagree |
| Strongly disagree |
| Comments: |
| Long answer text |
| Q20. What would you suggest to improve the impact of short term surgical missions? * |
| Long answer text |

| Q21. Hereby I give consent to use this data for publication. The purpose of this public provide more insight into short-term surgical missions | ation is to |
|---|---|
| ○ Yes | |
| ○ No | |